CLINICAL TRIAL: NCT00003060
Title: Pilot Study for Matched-Related Allogeneic Bone Marrow Transplantation for Metastatic Malignant Melanoma
Brief Title: Chemotherapy Plus Bone Marrow Transplantation in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of patient accrual
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: LSU-95456; CDR0000065722 (Registry Identifier: PDQ (Physician Data Query)); NCI-V97-1318
Record Dates: First submitted 1999-11-01; First posted 2003-11-25 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Clinical trial to study the effectiveness of chemotherapy plus bone marrow transplantation in treating patients with metastatic melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and survival of patients with metastatic malignant melanoma who have failed first-line therapy when treated with match-related allogeneic bone marrow transplantation.

OUTLINE: This is a pilot study. Patients receive a preparative regimen of busulfan and cyclophosphamide. Busulfan PO is administered every 6 hours on days -7 to -4. Cyclophosphamide IV is administered on days -3 to -2 followed by one day of rest. Bone marrow infusion occurs on day 0. Cyclosporine begins on day -1 and continues until day 180. Methotrexate IV is administered on days 1, 3, 6, and 11. Granulocyte colony-stimulating factor is administered as a continuous IV every 2 hours starting on day 12 and continuing until absolute neutrophil count is greater than 1,000 g/dL for 2 consecutive days. Patients receive weekly follow up for the first 180 days and monthly thereafter. Patients are followed until death.

PROJECTED ACCRUAL: 6 patients with melanoma will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy proven relapsed malignant melanoma that has failed prior standard regimen for metastatic disease Must have HLA-matched or related bone marrow donor (5- or 6-antigen match) No history of CNS metastases

PATIENT CHARACTERISTICS: Age: 16 to 44 Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: SGOT and SGPT less than 1.5 times upper limit of normal Bilirubin less than 1.5 mg/dL Renal: Creatinine less than 1.5 mg/dL AND/OR Creatinine clearance greater than 75 mL/min Cardiovascular: No history of cardiac disease No symptomatic cardiac disease Ejection fraction greater than 50% Pulmonary: FEV1 greater than 50% predicted (greater than 75% if received thoracic irradiation) DLCO greater than 50% predicted Other: Not pregnant Fertile women must use effective contraception HIV negative No active bacterial, fungal, or viral infection Hepatitis B negative

PRIOR CONCURRENT THERAPY: At least 1 prior standard regimen for metastatic disease

Ages: 16 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 1995-03; Primary Completion 2001-02-22 (Actual); Study Completion 2001-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin B. Weinberger, MD, Study Chair — Feist-Weiller Cancer Center at Louisiana State University Health Sciences
Locations (1):
- Louisiana State University School of Medicine, Shreveport, Louisiana, United States